CLINICAL TRIAL: NCT01531257
Title: Proteogenomic Monitoring and Assessment of Kidney Transplant Recipients
Acronym: Mini-Kidney
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Transplant Genomics, Inc. (Industry)
Responsible Party: Principal Investigator, Sook Hyeon Park, Assistant Professor of Medicine, Northwestern University
Other Study IDs: STU 25946
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Acute Rejection (AR) of Transplanted Kidney; Chronic Allograft Nephropathy (CAN); Interstitial Fibrosis (IF); Tubular Atrophy (TA)
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Collection: Approximately one cup of urine (200 mL) will be taken for research tests on the day of a routine care biopsy, if possible.
  Blood Draws: About 2.5 tablespoons of blood (38.5 mL) will be taken for research tests before the biopsy.
  Kidney Biopsy: A kidney biopsy is a procedure to remove and examine a small piece of kidney tissue. For this study, one biopsy will be taken from the new kidney and used specifically for research. The biopsy will be done at the same time as the biopsies done for routine care. If there are any complications during the routine care biopsies, the tissue for this research study will not be taken.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney Transplant Recipients: The intention of our biomarker panel is to be broadly applicable to all patients with a kidney transplant with the assumption that there are common underlying molecular mechanisms of AR and CAN/IFTA that can be detected hopefully at early stages of disease. We therefore want to validate and test our biomarker panel in a broad collection of patient types. We chose not to include patients with dual organ transplants so that we could isolate the molecular signal we are studying.

SUMMARY:
Chronic Allograft Nephropathy (CAN)/Interstitial fibrosis and Tubular Atrophy (IFTA) is responsible for most kidney transplant failures. CAN/IFTA on a 3 month kidney biopsy strongly predicts graft survival long term. CAN/IFTA remains a vexing problem for clinicians because current monitoring tools, namely the serum creatinine concentration, are not sensitive to early changes in glomerular filtration rate (GFR) or to histologic damage.

Despite advances in prevention of acute rejection (AR), it is still a significant and potentially devastating complication of solid organ transplantation. One strategy to reduce the risk of rejection is to perform kidney biopsies to detect subclinical acute rejection (SCAR) and treat to prevent progression to rejection. There is evidence that treating SCAR can prevent further immune mediated injury to the kidney, a precursor to CAN/IFTA.

Kidney biopsies provide better information but are limited due to safety concerns, patient preference and cost issues. Better, early and less invasive markers of CAN/IFTA will allow early intervention as well as improved graft and better patient outcomes.

This study seeks to validate specific proteogenomic biomarker panels for AR and CAN/IFTA in a prospective blood, urine and kidney tissue monitoring study of kidney transplant recipients who will be scheduled for standard of care biopsies.

DETAILED DESCRIPTION:
This is a single-center sample study. A total number of 1000 subjects will be consented and enrolled at Northwestern University Transplant clinic at the time of kidney biopsy. At our clinic, protocol biopsy may be performed at 3 months, 12 months , 24 months or any other time the doctor feels necessary post transplant in all kidney recipients. Kidney transplant recipients may also go under "for cause" biopsy procedure at any time point before/after or in between these protocol biopsy time points. Such causes of biopsy include increase in serum creatinine level, decrease in urine output, and/or pain at graft site.

Full blood tube set, urine sample for proteomics and flow cytometry of urinary sediment, and an extra core kidney biopsy tissue for gene expression profiling will be collected from subjects at the time of any biopsies obtained during the study course. These specimen samples will be sent to Rules-Based Medicine (RBM) for proteomic analysis. Whole genome expression profiling will be done using Affymetrix GeneChips at The Scripps Research Institute.

We estimate that we will find at least 500 subjects with diagnostic CAN/IFTA histology (Banff 1-2) between the 3 months and 12 months post transplant protocol biopsies based on a 50% incidence in the literature and our own experience. We also estimate that there will be 10% (10 subjects) incidence of clinical rejection by the end of 12 months identified initially by an acute rise in the serum creatinine and confirmed by a biopsy. Lastly, we estimate a 10% (10 subjects) incidence of subclinical acute rejection with stable renal function detected by the protocol kidney biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female recipients of all races, ≥18 years of age.
2. Patients undergoing primary or subsequent deceased-donor or living donor kidney transplantation.
3. Subject and/or guardian must be able to provide informed consent.
4. Subject and/or guardian must be able to comply with the study protocol.

Exclusion Criteria:

1. Need for combined organ transplantation with an extra-renal organ and/or islet cell transplant.
2. Recipients of previous non-renal solid organ and/or islet cell transplantation.
3. Infection with HIV.
4. Inability or unwillingness of a participant and/or guardian to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present for routine care kidney transplant biopsies to the Comprehensive Transplant Center and who satisfy all of the eligibility criteria are approached for this research study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-04; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Gene Expression Profiling | At time of any protocol or for-cause kidney biopsy, up to 10 years post transplant.
  Full blood tube set, urine sample for proteomics and flow cytometry of urinary sediment, and an extra core kidney biopsy tissue for gene expression profiling will be collected from subjects at the time of any biopsies obtained during the study course. Whole genome expression profiling will be done using Affymetrix GeneChips at The Scripps Research Institute.

CONTACTS AND LOCATIONS:
Overall Officials: Sook H Park, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States